CLINICAL TRIAL: NCT02195596
Title: Effects of Exercise on Cognitive Performance of Patients With Alzheimer-type Dementia. Pilot Study.
Acronym: EFA-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Ana Dosío Revenga, Family physician, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2011111100
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease, exercise, cognition
MeSH Terms: conditions — Alzheimer Disease; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High intensity aerobic exercise+strength (Experimental): The program consist in a "Continuous High aerobic exercise and moderate intensity intervals" (ShoshanaB et al, 2012) combined with "muscular strength exercises and joint mobility". Patients come three times a week for six months to the primary health center. A fitness expert nurse is responsible for monitoring the performance and adapt to the physical condition of the patient.Each exercise session consists of warming up time period, period of work and back to calm. Exercise intensity during the work period increases progressively as the program progresses. Aerobic exercise is performed on a cycle ergometer or treadmill.Muscle strength exercises and joint mobility are performed with dumbbells and ankle weights adapted to each patient.
  Interventions: Other: High intensity aerobic exercise+strength
- Low intensity aerobic exercise+strength (Active Comparator): The control group performed an exercise program similar to intervention but at low intensity that is below 35 or 40% of heart rate reserve (HRR).
  Interventions: Other: Low intensity aerobic exercise+strength

INTERVENTIONS:
Other: High intensity aerobic exercise+strength — The program consist in a "Continuous High aerobic exercise and moderate intensity intervals" (ShoshanaB et al, 2012) combined with "muscular strength exercises and joint mobility". Patients come three times a week for six months to the primary health center and will be supervised by an expert nurse.
  Arms: High intensity aerobic exercise+strength
Other: Low intensity aerobic exercise+strength — Low intensity aerobic exercise+strength program is similar to the other intervention but differs in the intensity of the exercise as it works with intensities below 40% of heart rate reserve.
  --------------------------------------------------------------------------------
  Arms: Low intensity aerobic exercise+strength

SUMMARY:
A program that combines high intensity aerobic exercise (<85% of Heart Rate Reserve) with resistance, progressive and moderate intensity intervals, carried out in primary care, is effective in terms of a smaller increase in respect to the baseline measurement in the total score of the ADAS cognitive section (Alzheimer Disease Assessment Scale-Cognitive section),in the control group that receives an intervention similar to low intensity (30-40% of Heart rate reserve).

We Expect a difference of at least 3 points between the means of the increments between the intervention and control group.

DETAILED DESCRIPTION:
OBJECTIVE: To evaluate an intervention that combines high intensity aerobic exercise with strength (AAAD) on general cognitive performance of patients affected by mild Alzheimer's disease (AD). DESIGN: Randomized clinical trial in two parallel groups: SCOPE: 2 health center of Basque Health Service , in coordination with its reference neurology services. PARTICIPANTS: 80 patients with mild AD.

INTERVENTION: Both groups receiving standard drug treatment. The intervention group also receive a supervised EEAA program, while the control group receive a similar intervention at low intensity. Patients are followed up over 1 year. Three blind measurements are made repeatedly : baseline, at 6 and 12 months. MEASUREMENTS: The primary outcome measure is change in cognitive performance that is measured in a blinded way with the cognitive section of the ADAS scale (Alzheimer's Disease Assessment Scale) at 0, 6 and 12.Secondary Outcomes: Global cognitive performance (Neuropsychological battery TBR-B),neuropsychiatric symptoms (NPI), ADL (Blessed),functional capacity (Test of 6-minute walk), cardiorespiratory Test, muscular strength (hand dynamometer and trunk); PREDICTORS AND CONFOUNDING VARIABLES: baseline cognitive performance, previous physical activity, medication, age, sex, APOE, schooling and cognitive reserve. ANALYSIS: We compared the two groups in terms of observed mean changes from baseline in ADAS measurement and other variables, intention to treat, using longitudinal mixed effects models for repeated measures at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria: Subjects aged between 55 and 85 who meet, at the time of entry into the study, clinical criteria compatible with probable AD according to the criteria of the National Institute on Aging and the Alzheimer's Association, under mild or DCL-Alzheimers (Folstein MMSE> 19/20, GDS 3-4), diagnosis will be performed by specialist neurologists according to standard practice. Patients should be able to perform physical activity on a cycle ergometer or treadmill and also must exist a caregiver who agrees to accompany him to the physical exercise sessions.

-

Exclusion Criteria: Central nervous system disease history with the possibility of neuropsychological impairment (stroke, epilepsy, meningitis, severe head trauma). History of alcohol and drug abuse. Hachinski Ischemic Scale ≥ 7. Major depression diagnosed(CIE-10). History of severe psychiatric disease. Predictable changes in medication that may affect cognitive performance. Visual or auditory perceptual disorders that limit neuropsychological assessment. Unstable heart disease, severe behavioral problems that make impossible the intervention, or any condition judged by the investigator that advises against the intervention. -

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-01 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive performance that is measured in a blinded way with the cognitive section of the ADAS scale (Alzheimer's Disease Assessment Scale) at 0, 6 and 12 | 0, 6 and 12 months
  Cognitive performance is measured in a blinded way with the cognitive section of the ADAS scale (Alzheimer's Disease Assessment Scale) at 0, 6 and 12. ADAS is an instrument designed to assess the severity of cognitive disorders (ADAS-Cog) and noncognitive (ADAS-cog) in patients with Alzheimer-type dementia (ATD). The ADAS-Cog, that we use, consists of 11 items that assess mainly memory (3 items, 27 points), orientation (1 item, 8 points), language (5 items, 25 points) and praxis (2 items, 10 points). The maximum score is 70 points.The higher the score, the greater the cognitive impairment.This is the primary outcome measure most frequently used in clinical trials with drugs.

SECONDARY OUTCOMES:
Global cognitive performance | 0, 6 and 12 months
  Global cognitive performance is measured with Test Barcelona TBR-B neuropsychological battery (abreviated version).The ADAS-COG wich is focused on the most devastated areas by Alzheimer's disease, will be complemented by the TBA-B, which has been developed in our environment, makes possible a more global assessment, and also presents adequate psychometric properties.

OTHER OUTCOMES:
neuropsychiatric symptoms and psychopathology | 0, 6 and 12 months
  NPI will be employed to asses treatment related behavioral changes and the presence of psychopathology in patients receiving exercise

CONTACTS AND LOCATIONS:
Overall Officials: ANA DOSIO REVENGA, PHD, Principal Investigator — Osakidetza
Locations (3):
- Spain (3):
  - Galdakao Hospital/Galdakao C.S., Galdakao, Bilbao
  - Basauri C.S., Basauri, Bizkaia
  - Hospital Universitario de Basurto, Bilbao, Bizkaia